CLINICAL TRIAL: NCT01377857
Title: HIV Screening Take-up: Evaluating Incentives and Opt-out Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10562983; 1RC4AG039078-01 (NIH)
Record Dates: First submitted 2011-06-18; First posted 2011-06-21 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Opt-In (Experimental): Opt-in refers to a default of no test - patients must ask for the test in order to receive it. Patients are informed of the availability of rapid testing. They are tested only if they request the test.
  Interventions: Behavioral: HIV Test Offering
- Opt-Out (Experimental): Opt-out has a default to test - patients are informed that they will receive a rapid HIV screening test unless they decline it. Patients will be tested unless they decline.
  Interventions: Behavioral: HIV Test Offering
- Active Choice (Experimental): In the active choice treatment, there is no default; patients must actively accept or actively decline the test.
  Interventions: Behavioral: HIV Test Offering
- $1 Incentive (Experimental): When offering the HIV test, study staff will inform subjects that the ED is offering cash incentives to promote HIV testing (and that the test is also free), and will inform them of that day's value.
  Interventions: Behavioral: Monetary Incentive
- $5 Incentive (Experimental): When offering the HIV test, study staff will inform subjects that the ED is offering cash incentives to promote HIV testing (and that the test is also free), and will inform them of that day's value.
  Interventions: Behavioral: Monetary Incentive
- $10 Incentive (Experimental): When offering the HIV test, study staff will inform subjects that the ED is offering cash incentives to promote HIV testing (and that the test is also free), and will inform them of that day's value.
  Interventions: Behavioral: Monetary Incentive
- Early Questionnaire (Experimental): At a time that does not interfere with patients' medical care, patients will be approached by a member of the research team to consent to and complete a short (3 minutes) questionnaire. The questionnaire is designed to elicit two things: subjective risk of infection (e.g., What are the chances you have HIV? [Not possible, Unlikely, Possible, Likely, Certain]) and objective risk of infection (e.g., In the past year, have you given anyone drugs or money for sex?). The questionnaire will be administered as one of two timing treatments - a) at the beginning of care, before the patient is offered an HIV test (Early questionnaire) or b) after the patient has been offered an HIV test (Late questionnaire).
  Interventions: Behavioral: Questionnaire Timing
- Late Questionnaire (Experimental): At a time that does not interfere with patients' medical care, patients will be approached by a member of the research team to consent to and complete a short (3 minutes) questionnaire. The questionnaire is designed to elicit two things: subjective risk of infection (e.g., What are the chances you have HIV? [Not possible, Unlikely, Possible, Likely, Certain]) and objective risk of infection (e.g., In the past year, have you given anyone drugs or money for sex?). The questionnaire will be administered as one of two timing treatments - a) at the beginning of care, before the patient is offered an HIV test (Early questionnaire) or b) after the patient has been offered an HIV test (Late questionnaire).
  Interventions: Behavioral: Questionnaire Timing
- FITD Questionnaire (Experimental): There will be two versions of the early questionnaire: one standard Early questionnaire, and one with an additional question: "If you were offered an HIV test as part of your routine health care at no cost, would you get tested?" The two questionnaires will be otherwise identical.
  Interventions: Behavioral: Questionnaire Timing
- Free (Experimental): When offering the HIV test, study staff will inform subjects that the ED is offering HIV testing (and that the test is also free); no monetary incentive will be offered.
  Interventions: Behavioral: Monetary Incentive

INTERVENTIONS:
Behavioral: Monetary Incentive — $1, $5, or $10 incentive
  Arms: $1 Incentive; $10 Incentive; $5 Incentive; Free
Behavioral: Questionnaire Timing — Timing of the questionnaire--either before or after testing is offered.
  Arms: Early Questionnaire; FITD Questionnaire; Late Questionnaire
Behavioral: HIV Test Offering — HIV Test will be offered as opt-in, opt-out, or active choice.
  Arms: Active Choice; Opt-In; Opt-Out

SUMMARY:
Over twenty percent of HIV-positive persons in the United States are unaware of their infection, leading the Institute of Medicine to recently urge further work to compare the effectiveness of HIV screening strategies. This study will use a randomized trial to compare several variants of emergency-room-based HIV-testing policies in order to determine how HIV test acceptance rates can be increased. The testing policies will be designed using principles from behavioral economics, varying the choice architecture and offering small monetary incentives. This will be the first study to measure differences in take-up rates across a variety of promising but largely untested approaches within a unified randomized trial. Three defaults will be tested: traditional opt-in (test only those patients who request testing), opt-out (routinely testing unless patients decline), and active-choice testing (patients are required to state whether they want to be tested). The study will also be the first to test the effect of small monetary incentives ($1, $5, $10) on test take-up. An additional novel study contribution will be to test the hypothesis that compliance with large requests (accept an HIV test) increases after making a small request or pre-commitment - this "foot in the door" technique has not been previously studied in this setting. The factorial design will permit a direct comparison of all interventions, as well as interactions. The study will contribute a nuanced empirical understanding of how testing protocols from behavioral economics theory affect the effectiveness and efficiency of screening programs in an actual scaled- up setting (San Francisco General Hospital). This will assist in implementing and assessing recent CDC guidelines on HIV screening, while also more generally advancing scientific knowledge related to applying behavioral economics in comparative effectiveness research.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 13 - 64 years who are awake, alert, not intoxicated, and understand the premise of the test will be offered the test and questionnaire according to their treatment group.

Exclusion Criteria:

* Patients who have altered levels of consciousness, are critically ill (e.g., serious trauma), are known to have preexisting HIV diagnosis, or who have been tested for HIV in the past 3 months will be excluded from the study.
* Pregnant patients will be excluded due to alternative guidelines for incorporating opt-out testing during prenatal care.
* Any patients who are in police custody will also be excluded due to their lack of control over study participation decisions and ethical concerns over possible coercion.

Ages: 13 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8572 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients offered an HIV test who accept | Monthly

SECONDARY OUTCOMES:
Proportion testing HIV positive of those tested | Monthly
Proportion testing HIV positive among those offered a test | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Beth Kaplan, MD, Principal Investigator — University of California, San Francisco; William H Dow, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Montoy JC, Dow WH, Kaplan BC. Patient choice in opt-in, active choice, and opt-out HIV screening: randomized clinical trial. BMJ. 2016 Jan 19;532:h6895. doi: 10.1136/bmj.h6895. PMID 26786744